CLINICAL TRIAL: NCT00517010
Title: Phase 1 Pilot Open Label Prospective Observational Study of Safety and Tolerability of Lucentis Combined With Proton Beam Irradiation in Treating Exudative Age-related Macular Degeneration
Brief Title: Pilot Study of Lucentis Combined With Proton Beam Irradiation in Treating Wet Age-related Macular Degeneration
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: University of California, San Francisco (Other); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200715285; 100,481 (Other: FDA IND)
Record Dates: First submitted 2007-08-15; First posted 2007-08-16 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-06

CONDITIONS: Age-related Macular Degeneration
Keywords: Age-related macular degeneration; Exudative age-related macular degeneration; Wet macular degeneration; Intravitreal injection; Proton beam irradiation; Lucentis; Ranibizumab
MeSH Terms: conditions — Macular Degeneration; Wet Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- proton beam with ranibizumab (Experimental): Intervention is 24Gy proton radiation in 2 fractions given within 6 weeks of first dose of intravitreal ranibizumab (0.5mg) drug combined with four monthly doses of intravitreal lucentis and monthly prn lucentis thereafter.
  Interventions: Drug: Proton beam irradiation and ranibizumab

INTERVENTIONS:
Drug: Proton beam irradiation and ranibizumab — ranibizumab 0.5mg intravitreal monthly x 4, then prn combined with low dose proton beam irradiation 24Gy (2 fractions, 24 hours apart) during the first month of study.
  Other Names: Lucentis and proton beam

SUMMARY:
Because a possible synergism of radiation and inhibitors of vascular endothelial growth factor has been shown in cancer patients and patients with wet macular degeneration, this pilot study is being conducted to determine whether treating wet macular degeneration with a combination of Lucentis and proton beam irradiation is safe. Lucentis is an inhibitor of vascular endothelial growth factor which was recently FDA approved for treatment of wet macular degeneration. It appears to be the most effective therapy thus far for wet macular degeneration among all drugs FDA approved for this condition. If no major safety issues are associated with this combination therapy, a larger study will be conducted to determine whether this combination therapy is more effective than Lucentis monotherapy.

DETAILED DESCRIPTION:
Five subjects diagnosed with wet macular degeneration will be treated with standard of care, i.e. intravitreal Lucentis injection monthly for the first four months and as needed thereafter. Within six weeks of the first Lucentis injection, the eye will also be treated with 24 Gy of proton beam divided into two fractions. Each subject will be followed for 2 yrs with monthly examination.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 50 years
* Patient related considerations
* Able to maintain follow-up for at least 24 months.
* Women must be postmenopausal without a period for at least one year.
* Hgb A1C < 6
* Diagnosed with Age-related Macular Degeneration (ARMD) with active subfoveal choroidal neovascular membrane (CNVM), new or recurrent
* Visual acuity 20/60 to 20/400
* Lesion size < 12 Disc Area
* Submacular hemorrhage less than 75% of total lesion
* Submacular fibrosis less than 25% of total lesion
* Candidate for intravitreal Lucentis

Exclusion Criteria:

* Prior enrollment in the study
* Pregnancy (positive pregnancy test) or lactation
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial
* CNVM within 1 mm from the disc margin
* Photodynamic Therapy (PDT) within 3 months
* Anti-VEGF therapy within 6 weeks
* Intravitreal or subtenon's Kenalog within 6 months
* Intraocular surgery within 3 months or expected in the next 6 months
* Current or planned participation in other experimental treatments for wet AMD
* Other concurrent retinopathy or optic neuropathy
* Other causes of CNVM, i.e. myopic degeneration or ocular histoplasmosis (POHS)
* Significant media opacity precluding adequate view of the fundus for exam,
* photography or OCT
* History of radiation therapy to the head or study eye
* Systemic anticoagulation with coumadin
* Head tremor or h/o claustrophobia precluding positioning for proton irradiation
* Inability to maintain steady fixation with either eye
* Diabetes mellitus requiring treatment
* History of Malignancy treated within 5 years
* Allergy to Fluorescein dye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanna S Park, MD PhD, Principal Investigator — University of California, Davis

IPD SHARING:
Plan to Share IPD: Yes
Findings have been presented at national and international venues and published in scientific peer-reviewed journal

REFERENCES:
- [Result] Park SS, Daftari I, Phillips T, Morse LS. Three-year follow-up of a pilot study of ranibizumab combined with proton beam irradiation as treatment for exudative age-related macular degeneration. Retina. 2012 May;32(5):956-66. doi: 10.1097/IAE.0b013e31822a8d6a. PMID 22183743

RESULTS

PARTICIPANT FLOW:
Groups:
- Lucentis Combined With Proton Beam: Proton beam irradiation and ranibizumab: ranibizumab 0.5mg intravitreal monthly x 4, then prn combined with low dose proton beam irradiation 24Gy (2 fractions, 24 hours apart) during the first month of study.
Period: Overall Study
Arm/Group | Lucentis Combined With Proton Beam
Started | 6
Completed | 5
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lucentis Combined With Proton Beam
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Best corrected visual acuity [Mean (Standard Deviation); unit: logMAR best corrected visual acuity] — Number of letters read correctly
  logMAR best corrected visual acuity | 0.58 (0.26)
Optical coherence tomography central macular thickness [Mean (Standard Deviation); unit: microns] — Central macular thickness for quantitative measure; qualitative measure of presence or absence of intraretinal or subretinal fluid
  microns | 335 (67)

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Ocular Adverse Events
Description: Any ocular adverse event identified by eye examination during the study follow-up will be recorded and determined for possible or probable relation to study treatment.
Time Frame: 24 months
Measure: Number; unit: number of adverse events
Arm/Group | Lucentis Combined With Proton Beam
Number analyzed (Participants) | 6
number of adverse events | 0

2. Secondary Outcome: 1. Change in BCVA From Baseline
Description: change in number of letter read correctly in study eye compared to the number of letters read correctly at baseline, i.e. BCVA (number of letters read correctly) at 24 months minus BCVA (number of letters read correctly) at baseline
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: change in number of letters
Arm/Group | Lucentis Combined With Proton Beam
Number analyzed (Participants) | 6
change in number of letters | 2.8 (26.4)

ADVERSE EVENTS:
Arm/Group | Lucentis Combined With Proton Beam
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No